CLINICAL TRIAL: NCT06630390
Title: Randomized, Double-blind Trial of Daridorexant to Prevent Delirium After Heart Surgery
Brief Title: Daridorexant to Prevent Delirium After Heart Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Mark Oldham, Associate Professor of Psychiatry, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00009841
Record Dates: First submitted 2024-09-30; First posted 2024-10-08 (Actual); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: POSTOPERATIVE DELIRIUM; POSTOPERATIVE COGNITIVE DECLINE
Keywords: delirium; sleep; cognitive decline; Alzheimer disease and related dementias
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications; Delirium; Cognitive Dysfunction; Alzheimer Disease | interventions — daridorexant

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the daridorexant or placebo arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daridorexant (Experimental): Oral daridorexant 50 mg (or 25 mg, if taking a moderate 3A4 inhibitor) each of the first three nights after heart surgery.
  Interventions: Drug: Daridorexant 50 mg
- Placebo (Placebo Comparator): Oral matching placebo each of the first three nights after heart surgery.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Daridorexant 50 mg — Administered consistent with labeling from the US Food and Drug Administration.
  Arms: Daridorexant
Other: Placebo — Identical appearing to daridorexant
  Arms: Placebo

SUMMARY:
The goal of this phase 2 clinical trial is to demonstrate the feasibility of the current study methods and obtain preliminary data for an adequately powered trial of daridorexant with the aim of preventing delirium after heart surgery. The main aims this feasibility trial aims to answer are to demonstrate: (1) the feasibility of study recruitment; (2) the ability deliver study compounds to subjects according to the proposed methods; and (3) completeness of data capture; and (4) recording of potential adverse events.

Participants will: (1) complete a baseline visit; (2) take the study drug--either daridorexant or placebo--each of the first 3 nights after heart surgery; and (3) be evaluated for sleep and delirium each of the first three days after heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* Having surgical aortic valve replacement or coronary artery bypass graft surgery at Strong Memorial Hospital
* Can provide informed consent
* Able to speak, read, and write English
* Family member or close friend available for collateral

Exclusion Criteria:

* Prior heart surgery
* Infectious endocarditis
* Emergency surgery
* Delirium at baseline
* Auditory/visual impairment preventing study procedures
* Active alcohol or substance misuse
* Psychotic disorder
* Dementia-level deficits
* Use of a sleep aid before surgery
* Use of a strong 3A4 inhibitor
* Intolerance to daridorexant
* Severe kidney or liver impairment
* Narcolepsy
* Any condition that, in the opinion of the PI, compromises patient safety or data quality if enrolled in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-02-16 (Actual); Study Completion 2025-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Oldham, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No
This trial is designed to demonstrate feasibility rather than test hypotheses of efficacy. As such, the data that will be obtained would be of very limited value if shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: IRB approval received on October 21, 2024, and the study was concluded on February 16, 2025 (date of last study evaluation).
Period: Overall Study
Arm/Group | Daridorexant | Placebo
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was closed after 11 subjects were enrolled as we had established feasibility.
Groups:
- Total: Total of all reporting groups
Arm/Group | Daridorexant | Placebo | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (2.9) | 69.6 (6.3) | 68.8 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 5 | 6 | 11
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA), version 8.1, provides a brief assessment of cognition. The total MoCA score ranges from 0 to 30, with lower scores indicating greater cognitive impairment. A total MoCA score less than 24 is consistent with mild cognitive impairment.
  units on a scale | 26 (2.4) | 25.8 (1.8) | 25.9 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Delirium
Description: In this feasibility trial, the primary outcome is rate of completion for delirium assessments--not whether patients developed delirium or the scores on delirium assessments. We aimed to evaluate subjects for delirium on each of the first three days after heart surgery using the Delirium Rating Scale, Revised-98, and the 3-minute Diagnostic Interview for the Confusion Assessment Method. Delirium based on DSM-5-TR diagnostic criteria would be diagnosed using the information from these two assessments. Below we report the number of subjects evaluated on each of the postoperative days.
Time Frame: First 3 days after surgery
Population: We attempted to perform delirium assessments for subjects on each of the 3 first days after surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Daridorexant | Placebo
Number analyzed (Participants) | 5 | 6
Participants
  Postoperative day 1 | 5 | 6
  Postoperative day 2 | 5 | 6
  Postoperative day 3 | 5 | 5

2. Secondary Outcome: Sleep Disturbance
Description: When evaluating subjects on each of the first 3 days after surgery, we ask subjects to rate their sleep on the preceding night using Richards-Campbell Sleep Questionnaire. This scale includes 6 items (sleep-related domains), each scored using a visual analog scale, ranging from 0 to 100. Higher scores indicate better sleep. Given that this is a feasibility study, we report the number of subjects evaluated for sleep on each of the postoperative days.
Time Frame: First 3 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Daridorexant | Placebo
Number analyzed (Participants) | 5 | 6
Participants
  Postoperative day 1 | 5 | 6
  Postoperative day 2 | 5 | 6
  Postoperative day 3 | 5 | 5

ADVERSE EVENTS:
Time Frame: We evaluate for potential adverse events on each of the first three postoperative days.
Arm/Group | Daridorexant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/6
Other Adverse Events (participants affected / at risk) | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daridorexant (N=5) | Placebo (N=6)
Subcortical stroke (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daridorexant (N=5) | Placebo (N=6)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Sleepiness (Nervous system disorders) | 5 (5) | 5 (5)
Fatigue (Nervous system disorders) | 5 (5) | 5 (5)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2025-02-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT06630390/Prot_000.pdf